CLINICAL TRIAL: NCT04797416
Title: The Evaluation of Consistency by Finger Stick Blood Glucose or Venous Blood Glucose of Flash Glucose Monitoring in Different Infiltration Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Professer, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020477
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes; Flash Glucose Monitoring; Conscience
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1-hour group (Active Comparator): The time between the activation of the sensor and the storage of the first blood glucose value is 1 hour.
  Interventions: Device: FGM infiltration 1 hour group
- 6-hour group (Experimental): The time between the activation of the sensor and the storage of the first blood glucose value is 6 hours.
  Interventions: Device: FGM infiltration 6-hour group
- 12-hour group (Experimental): The time between the activation of the sensor and the storage of the first blood glucose value is 12 hours.
  Interventions: Device: FGM infiltration 12-hour group

INTERVENTIONS:
Device: FGM infiltration 1 hour group — The sensor is activated immediately after wearing (including the time between the sensor activation and the first blood glucose value stored，about 1 hour).
  Arms: 1-hour group
Device: FGM infiltration 6-hour group — Reactivate the sensor 5 hours after wearing (including the time between the sensor activation and the first blood glucose value stored，about 1 hour).
  Arms: 6-hour group
Device: FGM infiltration 12-hour group — Reactivate the sensor 11 hours after wearing (including the time between the sensor activation and the first blood glucose value stored，about 1 hour).
  Arms: 12-hour group

SUMMARY:
This is a prospective randomized controlled study to evaluate consistency by finger stick blood glucose or venous blood glucose in different infiltration time (including the time between activation of the sensor and storage of the first blood glucose value) of Flash glucose monitoring(FGM). In this study, the relationship between the dynamic blood glucose and finger stick blood glucose or venous blood glucose in type 2 diabetes mellitus patients(T2DM), was explored. And the investigators also analyzed the deviation and accuracy of FGM in practical application,so as to provide a good reference for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes fit the 1999 who diagnostic criteria for diabetes
* Aged 18 or above
* Without serious complications, such as diabetic ketoacidosis, severe infection,severe cardiac insufficiency, severe liver and kidney diseases
* Voluntary and signed informed consent to participate
* Be able to read and understand Chinese, perform all research visits and tasks, and follow research instructions

Exclusion Criteria:

* Patients with known allergy to medical grade adhesive or isopropanol used for skin disinfection, edema, skin damage, scar, redness, infection, etc. during pregnancy or preparation of pregnancy or at the sensor application site (dorsal side of upper arm).
* The examinee took drugs such as ascorbic acid (vitamin C) and salicylic acid (an ingredient in aspirin and many painkillers) that affected the accuracy of the sensor.
* MRI is required during the study.
* The examinee had poor compliance and could not continue to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference value | Up to 21 days
  The difference between finger stick blood glucose or venous blood glucose and FGM value.

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China